CLINICAL TRIAL: NCT05051488
Title: Dynamic Decompressive Craniotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rohit Khanna, MD (Industry)
Collaborators: Halifax Health (Other)
Responsible Party: Sponsor-Investigator, Rohit Khanna, MD, Principal Investigator, NeuroVention, LLC
Organization: NeuroVention, LLC (Industry)
Other Study IDs: 1
Record Dates: First submitted 2021-09-03; First posted 2021-09-21 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Brain Edema; TBI (Traumatic Brain Injury); Stroke, Acute; Cerebral Hemorrhage; Brain Tumor
Keywords: decompressive craniotomy; dynamic craniotomy; craniectomy; cranial fixation plate; cerebral swelling; intracranial hypertension; cranioplasty
MeSH Terms: conditions — Brain Edema; Brain Injuries, Traumatic; Stroke; Cerebral Hemorrhage; Brain Neoplasms; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Dynamic craniotomy — Dynamic decompressive craniotomy with semi-rigid bone flap fixation
Device: Dynamic craniotomy — Dynamic decompressive craniotomy with semi-rigid bone flap fixation

SUMMARY:
Prospective observational study on patients undergoing decompressive craniotomy

DETAILED DESCRIPTION:
A prospective study of 20 neurosurgical patients evaluating the dynamic decompressive craniotomy technique using NeuroVention, LLC craniotomy bone flap fixation plates. The plates allow for rigid and semi-rigid bone flap fixation dependent on the implantation technique. A dynamic craniotomy involves bone flap fixation wherein a limited transient outward bone flap movement is allowed by the plates to compensate for an increase in intracranial pressure from brain swelling. The plates also prevent the craniotomy bone flap from sinking inside the skull and compressing on the brain. Cerebral decompression surgery is undertaken for patients with cerebral swelling from malignant strokes, medically intractable intracranial pressure elevation in traumatic brain injuries and brain tumors. The dynamic craniotomy technique eliminates or reduces the need for a cranioplasty surgery with a potentially significant improvement in outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing craniotomy who are at an increased risk for developing post- operative brain swelling or increased intracranial pressure from a malignant stroke
* Patients undergoing craniotomy who are at an increased risk for developing post- operative brain swelling or increased intracranial pressure from traumatic brain injury
* Patients undergoing craniotomy who are at an increased risk for developing post- operative brain swelling or increased intracranial pressure from brain tumors.

Exclusion Criteria:

* Patients with blown pupil (cerebral herniation),
* Massive brain swelling
* Dismal outcome not expected to survive more than 1-2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing craniotomy who are at an increased risk for developing post- operative brain swelling or increased intracranial pressure from malignant strokes, traumatic brain injury, and/or brain tumors. Patients not expected to survive will be excluded.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome | 6 months
  Modified Rankin Scale and Glasgow Outcome Score
Craniotomy bone flap healing | 3 months
  CT scan to assess rate of normal bone flap position

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khanna R, Ferrara L, Khanna S. Biomechanics of a novel reversibly expandable dynamic craniotomy bone flap fixation plate. J Neurosurg. 2019 Jan 4;132(2):560-567. doi: 10.3171/2018.8.JNS172614. Print 2020 Feb 1. PMID 30611148
- [Background] Khanna R, Ferrara L. Dynamic telescopic craniotomy: a cadaveric study of a novel device and technique. J Neurosurg. 2016 Sep;125(3):674-82. doi: 10.3171/2015.6.JNS15706. Epub 2015 Dec 11. PMID 26654180
- [Background] Khanna R. Dynamic Decompressive Craniotomy with a Novel Reversibly Expandable Plate. J Neurol Surg A Cent Eur Neurosurg. 2017 Jul;78(4):386-389. doi: 10.1055/s-0036-1594013. Epub 2016 Nov 30. PMID 27903020
- See also: Dynamic craniotomy video — http://vimeo.com/289289158